CLINICAL TRIAL: NCT02887729
Title: Analysis of Clinical and Molecular Genetic Data Influencing the Evolution and Response to Therapy of ADPKD Patients (Autosomal Dominant Polycystic Kidney Disease)
Acronym: GENKYST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: GENKYST
Record Dates: First submitted 2016-08-30; First posted 2016-09-02 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-08

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
Keywords: Polycystic disease
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood

SUMMARY:
Genkyst is a regional cohort involving up to nephrologists working in private and public nephrology centers in the West of France. It registers clinical and molecular genetic data of all consenting patients with ADPKD from this area.

ELIGIBILITY:
Inclusion Criteria:

* ADPKD patients followed in Nephrology centers in the West of France
* Age >17

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ADPKD patients followed in Nephrology centers in the West of France
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2010-06; Primary Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Clinical description of the patient | at the inclusion day

SECONDARY OUTCOMES:
Genetic analysis | at the inclusion day

CONTACTS AND LOCATIONS:
Overall Officials: Yannick Le Meur, MD PhD, Study Director — University Hospital, Brest
Locations (26):
- France (26):
  - AUB Brest, Brest, France
  - ECHO dialyse, Le Mans, France
  - CH Niort, Niort, France
  - ECHO Confluent, Rezé, France
  - CH de Saint Nazaire, Saint-Nazaire, France
  - CH Saint Malo, St-Malo, France
  - CHU Angers, Angers
  - CHU Brest, Brest
  - Centre Nephrologie et Dialyse d Armorique, Brest
  - CH La Roche Sur Yon, La Roche-sur-Yon
  - CH Le Mans, Le Mans
  - AUB Lorient, Lorient
  - CH Bretagne Sud, Lorient
  - AUB Morlaix, Morlaix
  - CHU Nantes, Nantes
  - CHU Poitiers, Poitiers
  - CH Centre Bretagne, Pontivy
  - AUB Quimper, Quimper
  - CHI de Cournouaille, Quimper
  - CHU Rennes, Rennes
  - Centre Heliomarin de Roscoff, Roscoff
  - CH Yves LE FOLL, Saint-Brieuc
  - ECHO Centre Ambulatoire, Saint-Herblain
  - CHU Tours, Tours
  - CH Bretagne Atlantique, Vannes
  - ECHO Vannes, Vannes